CLINICAL TRIAL: NCT02287779
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study to Assess the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Multiple Oral Doses of SHP626 in Overweight and Obese Adult Subjects
Brief Title: Safety and Tolerability Study of SHP626 in Overweight and Obese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHP626-101
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Non-Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — volixibat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SHP626 (Experimental): 9/12 subjects -1x daily dose of 20mg for 12 days 9/12 subjects-1x daily dose of 40mg for 12 days 9/12 subjects-1x daily dose of 80mg for 12 days 9/12 subjects-1x daily dose of 120mg for 12 days or dose lower than 80mg for 12 days 9/12 subjects-1x daily dose of 160mg for 12 days or dose lower than 80mg for 12 days 9/12 subjects-2x daily dose of SHP626 (dose TBD) for 12 days 9/12 subjects-2x daily dose of SHP626 (dose TBD; lower or higher than cohort 6) for 12 days 9/12 subjects-1x or 2x daily dose of SHP626 in an escalating titration (doses TBD). Initial 3 days of SHP626 followed by an increased dose of SHP626 for 3 days and finally a further increase in dose of SHP626 for 6 days 9/12 subjects will take a 1x or 2x daily dose of SHP626 in escalating titration (doses TBD; lower or higher dose than cohort 8). Initial 3 days of SHP626 followed by an increased dose of SHP626 for 3 days and finally a further increase in dose of SHP626 for 6 days
  Interventions: Drug: SHP626
- Placebo (Placebo Comparator): Three subjects per cohort will take a matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHP626
  Arms: SHP626
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will investigate the safety and tolerability of daily dosing regimens of SHP626 in overweight and obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Males that comply with any applicable contraceptive requirements or females of non-childbearing potential
* No history of active or chronic disease other than that allowed by study (hypertension, hyperlipidemia and GERD or heartburn)
* Has a body mass index of 25-35 kg/m2 with a body weight of greater than 140lbs (assessed at screening)

Exclusion Criteria:

* No history of alcohol or substance abuse, including use of tobacco
* No substantial changes in eating habits or exercise routine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2015-06-19 (Actual); Study Completion 2015-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (1):
- New Orleans Center for Clinical Research, Knoxville, Tennessee, United States

REFERENCES:
- [Derived] Palmer M, Jennings L, Silberg DG, Bliss C, Martin P. A randomised, double-blind, placebo-controlled phase 1 study of the safety, tolerability and pharmacodynamics of volixibat in overweight and obese but otherwise healthy adults: implications for treatment of non-alcoholic steatohepatitis. BMC Pharmacol Toxicol. 2018 Mar 16;19(1):10. doi: 10.1186/s40360-018-0200-y. PMID 29548345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at one study centre in North America, from 19 January 2015 to 19 June 2015.
Pre-assignment Details: Overall, 84 participants were randomised and completed the study.
Groups:
- Placebo: Participants received placebo matched to volixibat tablet orally for 12 days.
- Volixibat 5 mg BID: Participants received volixibat (SHP626) 5 milligram (mg) capsule orally twice a day (BID) for 12 days.
- Volixibat 10 mg QD: Participants received volixibat (SHP626) 10 mg capsule orally once a day (QD) for 12 days.
- Volixibat 20 mg QD: Participants received volixibat (SHP626) 20 mg capsule orally QD for 12 days.
- Volixibat 2-5-10-20 mg QD: Participants received volixibat (SHP626) 2 mg capsule orally QD on Days 1-3, 5 mg capsule orally QD on Days 4-6, 10 mg capsule QD orally on Days 7-9, and 20 mg capsule QD orally on Days 10-12.
- Volixibat 30 mg QD: Participants received volixibat (SHP626) 30 mg capsule orally QD for 12 days.
- Volixibat 40 mg QD: Participants received volixibat (SHP626) 40 mg capsule orally QD for 12 days.
- Volixibat 80-40-20 mg QD: Participants received volixibat (SHP626) 80 mg capsule orally QD on Day 1, 40 mg capsule orally QD on Day 2, and 20 mg capsule orally QD on Days 3-12.
Period: Overall Study
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Started | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Completed | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants for whom a randomization number was assigned and who had taken greater than equal (>=) 1 dose of investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD | Total
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 84
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 41.5 (9.47) | 37.1 (15.40) | 46.2 (7.61) | 33.3 (9.82) | 46.2 (7.82) | 44.6 (10.70) | 36.6 (8.92) | 33.2 (11.34) | 40.1 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 6
  Male | 18 | 9 | 7 | 9 | 9 | 8 | 9 | 9 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Standard Hematology
Description: TEAEs were defined as events that either had a start date on or after the first dose of investigational medicinal product (IMP) or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An adverse event (AE) that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE. Hematology parameters included evaluation of hemoglobin, hematocrit, red blood cells, platelets, white blood cell count; total and differential, neutrophils (absolute), eosinophils (absolute), monocytes (absolute), basophils (absolute) and lymphocytes (absolute).
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set included all participants for whom a randomization number was assigned and who had taken >= 1 dose of IMP.
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Fat Soluble Vitamins (Vitamin A, D, & E)
Description: TEAEs were defined as events that either had a start date on or after the first dose of IMP or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An AE that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE. Fat soluble vitamin included vitamin A (serum retinol), vitamin D (serum 25-hydroxycholecalciferol) and vitamin E (serum alfa-tocopherol).
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set.
Measure: Number; unit: participants
Groups:
- Volixibat 5 mg BID: Participants received volixibat (SHP626) 5 mg capsule orally BID for 12 days.
- Volixibat 10 mg QD: Participants received volixibat (SHP626) 10 mg capsule QD for 12 days.
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Lipid Panel
Description: TEAEs were defined as events that either had a start date on or after the first dose of IMP or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An AE that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE. Lipid panel parameters included evaluation of total cholesterol, triglycerides, high-density lipoprotein (HDL) cholesterol, very low-density lipoprotein (VLDL) cholesterol and low-density lipoprotein (LDL) cholesterol.
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set.
Measure: Number; unit: participants
Groups:
- Volixibat 10 mg QD: Participants received volixibat (SHP626) 10 mg capsule orally QD for 12 days.
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Thyroid Hormone Panel
Description: TEAEs were defined as events that either had a start date on or after the first dose of IMP or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An AE that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE. Thyroid hormone panel parameters included evaluation of thyroid hormones (TSH [thyroid stimulating hormone]; T3 [triiodothyronine] and T4 [thyroxine]).
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Coagulation
Description: TEAEs were defined as events that either had a start date on or after the first dose of IMP or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An AE that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE. Coagulation included international normalized ratio, activated partial thromboplastin time and prothrombin time.
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Standard Chemistry
Description: TEAEs were defined as events that either had a start date on or after the first dose of IMP or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An AE that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE. Standard chemistry parameters included evaluation of sodium, potassium, glucose, blood urea nitrogen, creatinine, calcium, chloride, thyrotropin, thyroxine, tri-iodothyronine, phosphorus, protein, bicarbonate or carbon dioxide, albumin, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyltransferase, alkaline phosphatase, total bilirubin, urate, beta-human chorionic gonadotropin and follicle-stimulating hormone levels. Participant with TEAE related to standard chemistry were reported with hepatic enzyme increase.
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Urinalysis Parameters
Description: TEAEs were defined as events that either had a start date on or after the first dose of IMP or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An AE that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE. Urinalysis parameters included evaluation of pH, glucose, protein, nitrites, leukocyte esterase, occult blood, ketones, bilirubin and specific gravity levels.
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Vital Signs
Description: TEAEs were defined as events that either had a start date on or after the first dose of IMP or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An AE that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE. Vital signs parameter included evaluation of orthostatic blood pressure, respiratory rate and body temperature.
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants
  Tachycardia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pyrexia | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Electrocardiogram (12-lead)
Description: TEAEs were defined as events that either had a start date on or after the first dose of IMP or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An AE that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE. Twelve lead electrocardiogram parameters [(heart rate (HR), PR, RR, QRS and QT intervals and information on T-wave morphology (normal/abnormal) and U-wave morphology (absent/normal or abnormal)] were assessed.
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Treatment-emergent Adverse Events (STEAEs)
Description: TEAEs were defined as events that either had a start date on or after the first dose of IMP or has a start date before the date of the first dose of IMP, but increased in severity on or after the date of the first dose of IMP. An AE that occurred more than 9 days after the date of the last dose of double-blind IMP was not counted as a TEAE.
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants
  Participants with TEAEs | 14 | 9 | 9 | 9 | 9 | 9 | 9 | 9
  Participants with STEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Who Discontinued From the Study
Description: as for outcome 10
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 21 | 9 | 9 | 9 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Average Total Fecal Bile Acid (FBA) Concentration
Description: Stool samples for the determination of total FBA were collected in 48-hour windows from 48 hours before dosing on Day 1 through Day 14. The average of daily total FBA excretion is calculated before (Day -1 and Day -2) as the first pre dose of IMP and after (Day 1-12) as the first post-dose of IMP. The FBA is calculated as Total FBA (micromoles) = FBA (micromol per liter) * weight (grams) divided by 10^3. Participants with fecal bile acid concentration and their average pre-first dose and average post-first dose were reported.
Time Frame: Day -2 up to Day 14
Population: Pharmacodynamic set consisted of all participant in the safety analysis set for whom the primary pharmacodynamic data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: nanomoles*gram per liter
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 20 | 8 | 9 | 9 | 9 | 9 | 8 | 9
nanomoles*gram per liter
  Average Pre First Dose | 183.84 (176.229) | 166.95 (84.057) | 172.49 (180.992) | 238.22 (211.406) | 364.78 (304.905) | 408.49 (475.553) | 335.89 (277.883) | 116.73 (91.962)
  Average Post First Dose | 224.75 (195.403) | 941.32 (338.783) | 668.64 (365.183) | 1051.86 (554.781) | 1055.60 (394.246) | 987.01 (321.184) | 1172.08 (591.774) | 665.82 (539.150)

13. Secondary Outcome: Mean Serum 7- Alpha-hydroxy-4-cholesten-3-one (C4) Concentration
Description: Serum 7- alpha-hydroxy-4-cholesten-3-one (C4) concentrations were reported.
Time Frame: Day -1 to Day 15
Population: Pharmacodynamic set.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 20 | 8 | 9 | 9 | 9 | 9 | 8 | 9
nanogram per milliliter
  Day -1, Pre-Dose | 15.702 (19.1363) | 10.956 (3.7149) | 13.806 (10.0637) | 11.129 (6.7566) | 19.549 (12.2775) | 24.726 (37.6474) | 47.138 (42.7980) | 22.632 (18.9895)
  Day -1, 5 Hours Post-Dose | 31.952 (29.6023) | 17.418 (9.3636) | 26.272 (24.6615) | 35.649 (22.7807) | 34.262 (19.5308) | 42.490 (37.9101) | 58.411 (61.0322) | 27.311 (14.7722)
  Day -1, 13 Hours Post-Dose | 11.830 (10.3028) | 6.224 (3.9307) | 10.463 (7.9914) | 15.812 (7.6084) | 17.013 (9.7056) | 16.459 (15.9875) | 26.676 (26.9306) | 13.977 (8.4524)
  Baseline | 17.464 (29.6114) | 10.644 (6.2617) | 10.441 (7.8955) | 15.446 (13.4289) | 26.871 (17.6706) | 25.269 (34.4194) | 45.714 (49.4616) | 19.453 (16.9595)
  Day 1, Pre-Dose | 17.464 (29.6114) | 10.644 (6.2617) | 10.441 (7.8955) | 15.446 (13.4289) | 26.871 (17.6706) | 25.269 (34.4194) | 45.714 (49.4616) | 19.453 (16.9595)
  Day 1, 5 Hours Post-Dose | 27.300 (21.4321) | 29.041 (18.4231) | 54.602 (47.7655) | 60.478 (22.8216) | 65.289 (22.8088) | 63.769 (54.1516) | 88.713 (53.8752) | 35.520 (18.2429)
  Day 1, 13 Hours Post-Dose | 22.930 (29.6148) | 32.991 (23.3494) | 57.611 (28.4635) | 60.922 (20.1868) | 65.478 (27.8476) | 88.300 (64.8546) | 104.150 (65.6060) | 66.311 (21.3091)
  Day 6, Pre-Dose | 34.048 (57.5519) | 100.788 (48.0025) | 103.789 (66.6396) | 114.289 (81.4964) | 157.718 (69.9298) | 134.378 (90.2305) | 190.025 (114.5808) | 111.346 (91.6773)
  Day 6, 5 Hours Post-Dose | 33.972 (20.7411) | 129.625 (71.4311) | 145.111 (84.6147) | 143.756 (80.3355) | 185.278 (88.4269) | 190.378 (96.9316) | 202.788 (122.4445) | 100.089 (45.3246)
  Day 6, 13 Hours Post-Dose | 15.847 (13.7638) | 71.200 (30.2892) | 84.611 (71.3102) | 88.722 (68.5693) | 98.122 (43.5820) | 110.167 (46.8967) | 129.100 (74.2770) | 76.811 (40.6780)
  Day 12, Pre-Dose | 23.299 (26.1217) | 97.538 (68.0330) | 101.522 (95.1932) | 118.900 (78.4954) | 198.311 (87.5824) | 169.778 (101.2574) | 192.225 (128.8916) | 107.200 (77.8666)
  Day 12, 5 Hours Post-Dose | 32.567 (24.7723) | 120.738 (61.5278) | 144.767 (130.3808) | 156.689 (67.9233) | 232.189 (106.7850) | 196.933 (118.2849) | 210.088 (117.8523) | 104.167 (68.2195)
  Day 12, 13 Hours Post-Dose | 16.497 (12.9150) | 77.636 (40.5962) | 80.189 (77.9001) | 90.400 (55.9921) | 152.989 (81.6364) | 114.500 (40.2073) | 107.875 (52.3505) | 66.444 (36.9048)
  Day 13, Pre-Dose | 21.822 (32.8831) | 130.750 (85.2496) | 84.544 (55.4006) | 85.822 (42.7988) | 184.222 (66.6179) | 126.322 (65.9867) | 128.738 (83.4282) | 72.867 (49.7977)
  Day 13, 5 Hours Post-Dose | 29.110 (22.6451) | 107.325 (59.7595) | 94.022 (73.9921) | 78.100 (34.5601) | 161.556 (95.9363) | 110.756 (49.6502) | 89.363 (39.2784) | 57.567 (28.0922)
  Day 13, 13 Hours Post-Dose | 22.728 (24.6379) | 67.660 (46.6124) | 53.333 (40.0821) | 65.833 (34.3484) | 78.911 (50.2001) | 66.633 (23.7029) | 66.550 (30.6498) | 50.333 (23.8917)
  Day 15, Pre-Dose | 21.848 (24.0679) | 14.454 (11.0078) | 25.908 (18.3102) | 19.906 (11.2784) | 38.434 (21.0173) | 38.870 (38.5249) | 37.300 (26.1975) | 17.563 (12.4113)
  Day 15, 5 Hours Post-Dose | 30.099 (19.2391) | 34.663 (14.0156) | 51.009 (39.8047) | 30.868 (19.5278) | 63.067 (34.0796) | 55.257 (47.2884) | 36.960 (18.2242) | 26.322 (12.8678)
  Day 15, 13 Hours Post-Dose | 19.140 (18.9237) | 21.068 (10.4419) | 31.759 (28.8913) | 23.667 (10.0772) | 49.867 (21.1864) | 29.282 (23.4813) | 32.750 (22.6428) | 19.173 (8.3821)

14. Secondary Outcome: Number of Participants With Stool Hardness Using Bristol Stool Chart
Description: Stool hardness was assessed after each evacuation using the bristol stool chart, a medical aid designed to classify the form of human feces into 7 categories where type 1 is the hardest and type 7 is the softest.
Time Frame: Day -2 to Day 14
Population: Pharmacodynamic set.
Measure: Number; unit: participants
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 20 | 8 | 9 | 9 | 9 | 9 | 8 | 9
participants
  Day -2: Type 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Day -2: Type 2 | 2 | 1 | 1 | 1 | 1 | 3 | 0 | 1
  Day -2: Type 3 | 5 | 3 | 1 | 1 | 3 | 1 | 1 | 1
  Day -2: Type 4 | 5 | 1 | 5 | 1 | 3 | 0 | 2 | 4
  Day -2: Type 5 | 3 | 0 | 1 | 3 | 0 | 1 | 1 | 1
  Day -2: Type 6 | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 0
  Day -2: Type 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Day -1: Type 1 | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 1
  Day -1: Type 2 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 2
  Day -1: Type 3 | 8 | 2 | 1 | 2 | 1 | 1 | 1 | 1
  Day -1: Type 4 | 3 | 1 | 4 | 1 | 3 | 3 | 3 | 1
  Day -1: Type 5 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Day -1: Type 6 | 3 | 1 | 1 | 1 | 1 | 2 | 2 | 0
  Day -1: Type 7 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Day 1: Type 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Day 1: Type 2 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 1
  Day 1: Type 3 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Day 1: Type 4 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Day 1: Type 5 | 1 | 4 | 1 | 2 | 1 | 0 | 0 | 1
  Day 1: Type 6 | 2 | 2 | 5 | 3 | 5 | 5 | 4 | 4
  Day 1: Type 7 | 1 | 1 | 2 | 4 | 0 | 2 | 3 | 1
  Day 2: Type 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 2: Type 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Day 2: Type 3 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 1
  Day 2: Type 4 | 5 | 1 | 1 | 0 | 0 | 1 | 1 | 0
  Day 2: Type 5 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1
  Day 2: Type 6 | 2 | 4 | 6 | 4 | 6 | 7 | 5 | 4
  Day 2: Type 7 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2
  Day 3: Type 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 3: Type 2 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Day 3: Type 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 3: Type 4 | 4 | 1 | 1 | 0 | 0 | 2 | 0 | 0
  Day 3: Type 5 | 3 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  Day 3: Type 6 | 1 | 4 | 5 | 8 | 4 | 7 | 4 | 7
  Day 3: Type 7 | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 1
  Day 4: Type 1 | 6 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 4: Type 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: Type 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Day 4: Type 4 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0
  Day 4: Type 5 | 3 | 1 | 3 | 1 | 0 | 1 | 0 | 0
  Day 4: Type 6 | 2 | 3 | 2 | 5 | 4 | 8 | 5 | 7
  Day 4: Type 7 | 0 | 1 | 0 | 2 | 3 | 0 | 2 | 1
  Day 5: Type 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5: Type 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5: Type 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 5: Type 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 5: Type 5 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Day 5: Type 6 | 4 | 5 | 6 | 5 | 6 | 5 | 5 | 8
  Day 5: Type 7 | 0 | 1 | 2 | 2 | 1 | 1 | 3 | 0
  Day 6: Type 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 6: Type 2 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 6: Type 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 6: Type 4 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0
  Day 6: Type 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Day 6: Type 6 | 4 | 4 | 4 | 7 | 7 | 6 | 3 | 7
  Day 6: Type 7 | 0 | 2 | 2 | 1 | 1 | 1 | 5 | 0
  Day 7: Type 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7: Type 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7: Type 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7: Type 4 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day 7: Type 5 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 1
  Day 7: Type 6 | 4 | 6 | 5 | 5 | 6 | 7 | 5 | 6
  Day 7: Type 7 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0
  Day 8: Type 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8: Type 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8: Type 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Day 8: Type 4 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 8: Type 5 | 2 | 2 | 3 | 0 | 2 | 1 | 1 | 0
  Day 8: Type 6 | 0 | 4 | 5 | 4 | 3 | 7 | 5 | 6
  Day 8: Type 7 | 1 | 0 | 0 | 3 | 2 | 1 | 2 | 1
  Day 9: Type 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 9: Type 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 9: Type 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 9: Type 4 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day 9: Type 5 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Day 9: Type 6 | 4 | 3 | 8 | 6 | 6 | 7 | 7 | 5
  Day 9: Type 7 | 0 | 2 | 0 | 3 | 1 | 1 | 1 | 2
  Day 10: Type 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: Type 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: Type 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: Type 4 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Day 10: Type 5 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Day 10: Type 6 | 1 | 5 | 4 | 4 | 7 | 8 | 3 | 5
  Day 10: Type 7 | 0 | 1 | 2 | 4 | 1 | 1 | 4 | 0
  Day 11: Type 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 11: Type 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 11: Type 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 11: Type 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 11: Type 5 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Day 11: Type 6 | 2 | 3 | 9 | 9 | 7 | 8 | 2 | 6
  Day 11: Type 7 | 0 | 4 | 0 | 0 | 1 | 1 | 5 | 1
  Day 12: Type 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day 12: Type 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 12: Type 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 12: Type 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 12: Type 5 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
  Day 12: Type 6 | 2 | 4 | 7 | 3 | 8 | 6 | 5 | 8
  Day 12: Type 7 | 0 | 1 | 0 | 4 | 0 | 1 | 3 | 0
  Day 13: Type 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 13: Type 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Day 13: Type 3 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
  Day 13: Type 4 | 6 | 0 | 1 | 2 | 2 | 0 | 2 | 0
  Day 13: Type 5 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Day 13: Type 6 | 4 | 2 | 3 | 1 | 2 | 0 | 3 | 1
  Day 13: Type 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14: Type 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Day 14: Type 2 | 5 | 1 | 0 | 0 | 2 | 3 | 1 | 4
  Day 14: Type 3 | 1 | 1 | 2 | 0 | 2 | 2 | 1 | 2
  Day 14: Type 4 | 3 | 3 | 2 | 4 | 3 | 3 | 2 | 1
  Day 14: Type 5 | 3 | 1 | 1 | 1 | 0 | 1 | 1 | 0
  Day 14: Type 6 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1
  Day 14: Type 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Volixibat
Time Frame: Day 1 to Day 14
Population: Pharmacokinetic set consisted of all participants in the safety analysis set for whom the primary pharmacokinetic data were considered sufficient and interpretable. Due to minimal absorption of volixibat no participant had sufficient and interpretable primary pharmacokinetic data.
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Volixibat (SHP626)
Time Frame: Day 1 to Day 14
Population: Pharmacokinetic set. Due to minimal absorption of volixibat no participant had sufficient and interpretable primary pharmacokinetic data.
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of the study drug administration up to 9 days after the last dose of study drug administration
Arm/Group | Placebo | Volixibat 5 mg BID | Volixibat 10 mg QD | Volixibat 20 mg QD | Volixibat 2-5-10-20 mg QD | Volixibat 30 mg QD | Volixibat 40 mg QD | Volixibat 80-40-20 mg QD
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 13/21 | 9/9 | 9/9 | 9/9 | 9/9 | 9/9 | 9/9 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Volixibat 5 mg BID (N=9) | Volixibat 10 mg QD (N=9) | Volixibat 20 mg QD (N=9) | Volixibat 2-5-10-20 mg QD (N=9) | Volixibat 30 mg QD (N=9) | Volixibat 40 mg QD (N=9) | Volixibat 80-40-20 mg QD (N=9)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (27) | 9 (33) | 9 (27) | 9 (32) | 9 (26) | 9 (16) | 9 (26) | 9 (22)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
None of the participants in the safety analysis set were included in the pharmacokinetic set because no participant had sufficient and interpretable primary pharmacokinetic data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.